CLINICAL TRIAL: NCT00277641
Title: Lamotrigine in the Treatment of Binge Eating Disorder Associated With Obesity: A Single-Center, Double-Blind, Placebo-Controlled, Flexible-Dose Study in Outpatients
Brief Title: Lamotrigine in the Treatment of Binge Eating Disorder Associated With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: GlaxoSmithKline (Industry); University of Cincinnati (Other)
Responsible Party: Susan L. McElroy, MD, University of Cincinnati & Lindner Center of HOPE
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 106531
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: Binge Eating Disorder Associated with Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): lamotrigine
  Interventions: Drug: Lamotrigine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lamotrigine — 25 mg or 100 mg
  Arms: 1
Drug: placebo — identical tablets to study drug
  Arms: 2

SUMMARY:
This research study is to evaluate the effectiveness, tolerability, and safety of lamotrigine therapy in the treatment of binge eating disorder associated with obesity.

Lamotrigine has been approved by the Food and Drug Administration for the treatment of bipolar disorder, but has not been approved for use in the treatment of binge eating disorder with obesity.

DETAILED DESCRIPTION:
This is a 17-week, parallel group, placebo-controlled, randomized, double-blind, flexible-dose, single-center study. It begins with a 1 to 2 week screening period during which there will be washout of other medications and evaluation of protocol-specified criteria. The screening period will consist of at least two visits, which will include the initial screening visit and the baseline (week 1) visit. The treatment period follows the screening period and will last 16 weeks. Once a subject enters the treatment phase (after randomization) the dosage of study medication will be 25 mg/qHS (or one placebo tablet at night) for 14 days. On day 14 (visit 2 or the beginning of week 3), the dosage will be increased, as tolerated, to 25 mg b.i.d. On day 28 (visit 4 or in the beginning of week 5), the dosage will be increased, as tolerated, to 50 mg b.i.d. On day 35 (visit 5 or the beginning of week 6), the dosage will be increased, as tolerated, to 100 mg b.i.d. The dosage may be decreased at any time because of side effects. If the patient prefers, he or she may take all of his or her daily dose of medication in the morning or evening. If no response or an inadequate response (< 50% reduction in binge eating episodes compared with baseline) is evident by week 6 (visit 6), study medication may be increased to 150 mg b.i.d. If no response or an inadequate response is evident by week 8 (visit 7), study medication may be increased to 200 mg b.i.d. During weeks 12 through 16 (maintenance period) the dosage will not be changed unless a medical reason (e.g., adverse effect) requires such a change. The minimum dosage allowed will be 50 mg/day and the maximum dosage allowed will be 400 mg/day. The 16-week treatment period will be followed by medication discontinuation and evaluation 1 week after medication discontinuation (week 17). Efficacy and safety evaluations will be done at each visit starting with the baseline visit through week 17 (baseline, weeks 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16).

ELIGIBILITY:
Inclusion Criteria:

* Patients will meet DSM-IV-TR criteria for BED for at least the last 6 months, determined by the Structured Clinical Interview for DSM-IV-TR (SCID) (61) and supported by the Eating Disorder Examination (EDE) (62). These criteria are as follows:

  * Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following:

    * eating, in discrete period of time (e.g., within any two hour period), an amount of food that is definitely larger than most people would eat in a similar period of time under similar circumstances
    * a sense of lack of control over eating during the episode (e.g., a feeling that one cannot stop eating or control what or how much one is eating)
  * The binge eating episodes are associated with at least three of the following:

    * eating much more rapidly than normal
    * eating until uncomfortably full
    * eating large amounts of food when not feeling physically hungry
    * eating alone because of being embarrassed by how much one is eating
    * feeling disgusted with oneself, depressed, or feeling very guilty after overeating
  * Marked distress regarding binge eating.
  * The binge eating occurs, on average, at least two days a week for six months.
  * Does not occur exclusively during the course of bulimia nervosa and anorexia nervosa.
* Obesity, defined by body mass index > 30 kg/m2.
* Men or women, between the ages of 18 and 65.

Exclusion Criteria:

* Have current body mass index < 30 kg/m2.
* Women who are pregnant or lactating and women of childbearing potential who are not taking adequate contraceptive measures. (All women of childbearing potential will have a negative pregnancy test before entering the study.)
* Subjects who are displaying clinically significant suicidality or homicidality.
* Subjects who are displaying a current clinically unstable depressive or bipolar disorder, defined as a Montgomery Asberg Depression Rating Scale (MADRS) (63) > 24 or a Young Mania Rating Scale (YMRS) (64) > 8.
* A current or recent (within 6 months of the start of study medication) DSM-IV-TR diagnosis of substance abuse or dependence.
* A lifetime history of a DSM-IV-TR psychotic disorder or dementia.
* History of a personality disorder (e.g., schizotypal, borderline, or antisocial) which might interfere with assessment or compliance with study procedures.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, assessment, or treatment of binge eating disorder. Patients should be biochemically euthyroid prior to entering the study.
* History of seizures, including febrile seizures in childhood.
* Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication (e.g., stimulants, sympathomimetics, antidepressants, carbonic anhydrase inhibitors, anti-obesity drugs).
* Subjects who have received psychoactive medication (other than zaleplon [Sonata] or zolpidem [Ambien] -- as needed for restlessness/insomnia) within one week prior to randomization.
* Subjects who have begun and/or are receiving formal psychotherapy (cognitive behavioral therapy, interpersonal therapy, or dietary behavioral therapy) for BED or weight loss within the past 3 months.
* Subjects previously enrolled in this study or have previously been treated with lamotrigine.
* Subjects who have received an experimental drug or used an experimental device within 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The specific aims of this study are to examine the efficacy and safety of lamotrigine compared with placebo in outpatients with binge eating disorder associated with obesity. | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McElroy, MD, Principal Investigator — Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] Guerdjikova AI, McElroy SL, Welge JA, Nelson E, Keck PE, Hudson JI. Lamotrigine in the treatment of binge-eating disorder with obesity: a randomized, placebo-controlled monotherapy trial. Int Clin Psychopharmacol. 2009 May;24(3):150-8. doi: 10.1097/YIC.0b013e328329c7b5. PMID 19357528